CLINICAL TRIAL: NCT07390500
Title: Randomized Controlled Double Masked, Trial to Assess the Efficacy and Safety of a DYnaMic Peripheral DegradatiON Myopia Disorder Control in Myopic Children Compared to No Treatment (DYMOND Study)
Brief Title: Assessment of the Efficacy and Safety of a DYnaMic Peripheral DegradatiON Myopia Disorder Control in Myopic Children ״DYMOND Study״
Acronym: DYMOND
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: NovaSight (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NS-01317
Record Dates: First submitted 2026-01-29; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Myopia
Keywords: Myopia, myopia control, TrackSight, real-time eye-tracking technology
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants, parents, investigators, and study staff do not know whether the active visual feature is enabled.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- TrackSight™ with active peripheral image degradation (blur) (Experimental): Participants use TrackSight™ with active peripheral image degradation enabled using combination #1 during their normal screen activities. Central vision remains clear while the peripheral image is digitally modified. Standard single-vision glasses are worn at all times.
  Interventions: Device: TrackSight
- rackSight™ with active peripheral image degradation (contrast) (Experimental): Participants use TrackSight™ with active peripheral image degradation enabled using combination #2, which applies a different level or pattern of visual modification during screen use. Central vision is unaffected, and standard single-vision glasses are worn throughout the study.
  Interventions: Device: TrackSight
- TrackSight™ with the peripheral image degradation function disabled (control). (Sham Comparator): Participants use the same TrackSight™ software and device, but the peripheral image degradation feature is disabled. Screen use and standard single-vision glasses remain unchanged, serving as the control condition.
  Interventions: Device: TrackSight

INTERVENTIONS:
Device: TrackSight — applying a predefined combination of peripheral chromatic blur and contrast reduction during normal screen use

SUMMARY:
The DYMOND study evaluates the safety and effectiveness of TrackSight™, a digital medical application designed to slow myopia (nearsightedness) progression in children during everyday screen use. TrackSight uses eye-tracking technology to keep central vision clear while subtly adjusting the image in the peripheral viewing area, based on established scientific principles known to influence eye growth.

Up to 150 children aged 6 to 12 with myopia will participate at sites in Israel and Hong Kong. All participants will continue wearing their regular single-vision glasses and will be randomly assigned to use TrackSight with or without active visual adjustment for 12 months. Eye examinations and safety assessments will be conducted at the start of the study and after 6 and 12 months. The study aims to determine whether this non-invasive digital approach can safely slow myopia progression in children.

DETAILED DESCRIPTION:
The DYMOND study is a clinical research study designed to evaluate the safety and effectiveness of a digital application called TrackSight™ for slowing the progression of myopia (nearsightedness) in children. Myopia often worsens during childhood, particularly during activities that involve prolonged screen use, such as studying, gaming, or watching videos. This study explores whether a software-based approach can help reduce the rate of myopia progression during everyday screen use.

TrackSight™ is a software medical device that uses real-time eye-tracking technology to subtly adjust the visual information presented on a digital screen. While central vision remains clear at all times, the software applies controlled visual changes to the peripheral areas of the screen. These changes are designed to influence how the eye grows, based on established scientific principles that have been shown to slow myopia progression in studies using special spectacle and contact lenses. TrackSight delivers these same principles digitally, without altering standard vision correction.

Up to 150 children between the ages of 6 and 12 with mild to moderate myopia will participate in the study at clinical sites in Israel and Hong Kong. All children will continue wearing their regular single-vision glasses throughout the study. Participants will be randomly assigned to one of three study groups. Two groups will use TrackSight with different active visual adjustment settings, while one group will use the same application with these features turned off. Neither the families nor the study staff will know which version of the software a child is using during the study.

Children will use the TrackSight application during their normal screen activities over a period of 12 months. Eye examinations will be performed at the start of the study and again at 6 and 12 months to measure changes in eye growth and vision. Questionnaires will be used to assess screen use, vision-related quality of life, and overall experience with the software. Safety will be closely monitored throughout the study, and families will have access to technical support if needed.

The primary goal of the study is to determine whether TrackSight can safely slow the progression of myopia by reducing eye growth over one year compared with no active treatment. The results of this study may help support a new, non-invasive digital approach to managing childhood myopia in modern screen-based environments.

ELIGIBILITY:
Inclusion Criteria:

* Aged 6-12 years

  -. Diagnosed with myopia: cycloplegic spherical or spherical equivalent (SER) between -0.75D and -5.00D, astigmatism ≤ -1.50D, anisometropia < 1.50D
* Visual acuity 20/32 or better (age-appropriate testing) in both eyes
* Interocular VA difference ≤1.00 logMAR line
* Subject in general good health and able, as per investigator decision, to comply with study visits and protocol procedures
* The subject is using digital devices for at least 1 hour/day regularly according to parental report
* Signed informed consent by legal parent/guardian and assent approval -. Currently wearing single vision refractive correction

Exclusion Criteria:

* Past or concurrent use of any other myopia treatment (e.g., atropine, orthokeratology, myopia control glasses/lenses)
* Eye diseases or abnormality, developmental conditions, or past ocular surgeries or any other condition which could potentially affect refraction or AL progression according to the investigator's judgement
* Current or prior history of manifest strabismus, amblyopia, or nystagmus
* Subject cannot pass eye tracking calibration in at least 50% of cases, or cannot be tracked in at least 50% of the time during a screening eligibility test
* Current or previous use of bifocal lenses, progressive-addition lenses, or multi-focal contact lenses
* Premature gestational age ≤32 weeks or birth weight <1500g.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2025-12-24 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
change in axial length | 12 months
  change in axial length (AL) of the eye used to assess whether TrackSight™ slows eye growth compared with the control condition.

CONTACTS AND LOCATIONS:
Locations (1):
- Kaplan MC, Rehovot, Israel

IPD SHARING:
Plan to Share IPD: No
private sponsor study